CLINICAL TRIAL: NCT04481204
Title: PIONEER-Panc: Phase II Investigations of New and Emerging Therapies for Pancreatic Cancer
Brief Title: New and Emerging Therapies for the Treatment of Resectable, Borderline Resectable, or Locally Advanced Pancreatic Cancer, PIONEER-Panc Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0075; NCI-2020-04886 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0075 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Borderline Resectable Pancreatic Adenocarcinoma; Locally Advanced Pancreatic Ductal Adenocarcinoma; Resectable Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorouracil; dehydroftorafur; Gemcitabine; Irinotecan; Leucovorin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Oxaliplatin; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Control arm GroupI(mFOLFIRINOX) (Active Comparator): Patients receive mFOLFIRINOX for 3 months before and after surgery in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan; Drug: Leucovorin; Drug: Oxaliplatin
- Control arm GroupII(chemotherapy, FOLFIRINOX) (Active Comparator): Patients receive gemcitabine, gemcitabine and nab-paclitaxel, gemcitabine and cisplatin, or FOLFIRINOX for up to 4 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Drug: Gemcitabine; Drug: Irinotecan; Drug: Leucovorin; Drug: Nab-paclitaxel; Drug: Oxaliplatin
- Control arm GroupIII(FOLFIRINOX, radiation therapy) (Active Comparator): Patients receive FOLFIRINOX for 4-6 months in the absence of disease progression or unacceptable toxicity. Patients may then undergo radiation therapy at the discretion of medical doctors.
  Interventions: Drug: Fluorouracil; Drug: Irinotecan; Drug: Leucovorin; Drug: Oxaliplatin; Radiation: Radiation Therapy
- Control arm GroupIV(chemotherapy,FOLFIRINOX,radiation therapy) (Active Comparator): Patients receive gemcitabine, gemcitabine and nab-paclitaxel, gemcitabine and cisplatin, or FOLFIRINOX for 6 months in the absence of disease progression or unacceptable toxicity. Patients may then undergo radiation therapy at the discretion of medical doctors.
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Drug: Gemcitabine; Drug: Irinotecan; Drug: Leucovorin; Drug: Nab-paclitaxel; Drug: Oxaliplatin; Radiation: Radiation Therapy
- Control arm GroupV(FOLFIRINOX, radiation therapy) (Active Comparator): Patients receive FOLFIRINOX for 4-6 months in the absence of disease progression or unacceptable toxicity. Patients may then undergo radiation therapy at the discretion of medical doctors
  Interventions: Drug: Fluorouracil; Drug: Irinotecan; Drug: Leucovorin; Drug: Oxaliplatin; Radiation: Radiation Therapy
- Control arm GroupVI(chemotherapy,FOLFIRINOX,radiation therapy) (Active Comparator): Patients receive gemcitabine, gemcitabine and nab-paclitaxel, gemcitabine and cisplatin, or FOLFIRINOX for 6 months in the absence of disease progression or unacceptable toxicity. Patients may then undergo radiation therapy at the discretion of medical doctors
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Drug: Gemcitabine; Drug: Irinotecan; Drug: Leucovorin; Drug: Nab-paclitaxel; Drug: Oxaliplatin; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Control arm GroupII(chemotherapy, FOLFIRINOX); Control arm GroupIV(chemotherapy,FOLFIRINOX,radiation therapy); Control arm GroupVI(chemotherapy,FOLFIRINOX,radiation therapy)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
  Arms: Control arm GroupII(chemotherapy, FOLFIRINOX); Control arm GroupIV(chemotherapy,FOLFIRINOX,radiation therapy); Control arm GroupVI(chemotherapy,FOLFIRINOX,radiation therapy)
Drug: Irinotecan — Given IV
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
  Arms: Control arm GroupII(chemotherapy, FOLFIRINOX); Control arm GroupIV(chemotherapy,FOLFIRINOX,radiation therapy); Control arm GroupVI(chemotherapy,FOLFIRINOX,radiation therapy)
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Control arm GroupIII(FOLFIRINOX, radiation therapy); Control arm GroupIV(chemotherapy,FOLFIRINOX,radiation therapy); Control arm GroupV(FOLFIRINOX, radiation therapy); Control arm GroupVI(chemotherapy,FOLFIRINOX,radiation therapy)

SUMMARY:
This is a phase II study using the Bayesian platform design. There are three clinical stage groups of localized pancreatic cancer: resectable, borderline resectable, and locally advanced disease. Each stage group will have a defined standard of care chemotherapy regimen for a control arm, serving as a basis of comparison. Each group may have one or more experimental arms. Experimental arms may be added to the platform over time, and the effects of the experimental treatments will be tested against the controls for each group.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate major pathological response rate. (Resectable and borderline resectable groups [treatment naive or previously treated]) II. To estimate 6-month disease control rate. (Locally advanced groups [treatment naive or previously treated])

SECONDARY OBJECTIVES:

I. To measure progression free survival and overall survival. (Resectable and borderline resectable groups [treatment naive or previously treated]) II. To measure progression free survival and overall survival. (Locally advanced groups [treatment naive or previously treated])

EXPLORATORY OBJECTIVES:

I. To benchmark tissue acquisition protocols for deoxyribonucleic acid (DNA) and ribonucleic acid (RNA) analysis in pancreatic ductal adenocarcinoma (PDAC).

II. To demonstrate concordance of cell free DNA detected mutations to those detected in the tumor-derived DNA in PDAC.

III. To demonstrate response through exosome and circulating tumor DNA. IV. To demonstrate response through the quantification of the immune activation by analyzing T and B cells, peripheral blood mononuclear cells, and tissue biopsies.

V. To derive organoids from human PDAC and measure drug response in vitro. VI. To analyze the tumor microenvironment through immunohistochemistry (IHC) and hypoxia staining.

VII. To associate prognosis of patients with baseline and follow-up quantitative computed tomography (CT) image based analysis.

VIII. To associate clinical and pathological outcomes of patients with changes in radiomic measurements.

IX. To correlate quality of life for patients on standard and experimental therapies with laboratory, radiological, pathological, and clinical characteristics.

OUTLINE:Patients are assigned to different groups, and each group has a control arm. Within each group, the patient will be randomized to the appropriate control or an experimental arm. The control arms for the groups are:

Control arm for Group I (Treatment-naive resectable PDAC): Patients receive fluorouracil, irinotecan, leucovorin, and oxaliplatin (mFOLFIRINOX) for 3 months before and after surgery in the absence of disease progression or unacceptable toxicity.

Control arm for Group II (Previously-treated resectable PDAC): Patients receive gemcitabine, gemcitabine and nab-paclitaxel, gemcitabine and cisplatin, or FOLFIRINOX for up to 4 months in the absence of disease progression or unacceptable toxicity.

Control arm for Group III (Treatment-naive borderline resectable PDAC): Patients receive FOLFIRINOX for 4-6 months in the absence of disease progression or unacceptable toxicity. Patients may then undergo radiation therapy at the discretion of medical doctors.

Control arm for Group IV (Previously-treated borderline resectable PDAC): Patients receive gemcitabine, gemcitabine and nab-paclitaxel, gemcitabine and cisplatin, or FOLFIRINOX for 6 months in the absence of disease progression or unacceptable toxicity. Patients may then undergo radiation therapy at the discretion of medical doctors.

Control arm for Group V (Treatment-naive locally advanced PDAC): Patients receive FOLFIRINOX for 4-6 months in the absence of disease progression or unacceptable toxicity. Patients may then undergo radiation therapy at the discretion of medical doctors.

Control arm for Group VI (Previously-treated locally advanced PDAC): Patients receive gemcitabine, gemcitabine and nab-paclitaxel, gemcitabine and cisplatin, or FOLFIRINOX for 6 months in the absence of disease progression or unacceptable toxicity. Patients may then undergo radiation therapy at the discretion of medical doctors.

After completion of study treatment, patients are followed up every 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* TREATMENT NAIVE RESECTABLE PDAC COHORT: Pathologically proven adenocarcinoma of the pancreas by cytology or biopsy
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Confirmation of clinical stage of resectable
* TREATMENT NAIVE RESECTABLE PDAC COHORT: No prior chemotherapy or radiation therapy for PDAC
* TREATMENT NAIVE RESECTABLE PDAC COHORT: No current use of immunosuppressive medication
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Not pregnant and not nursing, for women of childbearing potential, a negative urine or blood pregnancy test done =< 7 days prior to registration is required
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Life expectancy greater than 6 months
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Absolute neutrophil count (ANC) >= 1,500/mm^3
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Platelet count >= 100,000/mm^3
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Creatinine =< 1.5 x upper limit of normal (ULN)
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Calculated (Calc.) creatinine clearance > 45 mL/min
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Total bilirubin =< 2.0 mg/dL
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Hemoglobin >= 8.0 mg/dL
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Pathologically proven adenocarcinoma of the pancreas by cytology or biopsy
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Confirmation of clinical stage of resectable
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Prior chemotherapy for PDAC is allowed, as long as the regimen is considered a standard regimen for PDAC (e.g., gemcitabine, gemcitabine-cisplatin, gemcitabine/nab-paclitaxel, gemcitabine/capecitabine, FOLFIRINOX). This should be discussed with the study principal investigators (PIs) prior to enrollment to ensure the regimen for a given patient is acceptable
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: No current use of immunosuppressive medication
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Not pregnant and not nursing, For women of childbearing potential, a negative urine or blood pregnancy test done ≤ 7 days prior to registration is required
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Life expectancy greater than 6 months
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: ECOG performance status 0 or 1
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Absolute neutrophil count (ANC) >= 1,500/mm^3
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Platelet count >= 100,000/mm^3
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Creatinine =< 1.5 x upper limit of normal (ULN)
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Calc. creatinine clearance > 45 mL/min
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Total bilirubin =< 2.0 mg/dL
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: AST/ALT =< 2.5 x upper limit of normal (ULN)
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Hemoglobin >= 8.0 mg/dL
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Pathologically proven adenocarcinoma of the pancreas by cytology or biopsy
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Confirmation of clinical stage of borderline resectable
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: No prior chemotherapy or radiation therapy for PDAC
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: No current use of immunosuppressive medication
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Not pregnant and not nursing, For women of childbearing potential, a negative urine or blood pregnancy test done ≤ 7 days prior to registration is required
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Life expectancy greater than 6 months
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: ECOG performance status 0 or 1
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Absolute neutrophil count (ANC) >= 1,500/mm^3
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Platelet count >= 100,000/mm^3
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Creatinine =< 1.5 x upper limit of normal (ULN)
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Calc. creatinine clearance > 45 mL/min
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Total bilirubin =< 2.0 mg/dL
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: AST/ALT =< 2.5 x upper limit of normal (ULN)
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Hemoglobin >= 8.0 mg/dL
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Pathologically proven adenocarcinoma of the pancreas by cytology or biopsy
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Confirmation of clinical stage of borderline resectable
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Prior chemotherapy for PDAC is allowed, as long as the regimen is considered a standard regimen for PDAC (e.g., gemcitabine, gemcitabine-cisplatin, gemcitabine/nab-paclitaxel, gemcitabine/capecitabine, FOLFIRINOX). This should be discussed with the study PIs prior to enrollment to ensure the regimen for a given patient is acceptable
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: No current use of immunosuppressive medication
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Not pregnant and not nursing, For women of childbearing potential, a negative urine or blood pregnancy test done =< 7 days prior to registration is required
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Life expectancy greater than 6 months
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: ECOG performance status 0 or 1
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Absolute neutrophil count (ANC) >= 1,500/mm^3
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Platelet count >= 100,000/mm^3
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Creatinine =< 1.5 x upper limit of normal (ULN)
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Calc. creatinine clearance > 45 mL/min
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Total bilirubin =< 2.0 mg/dL
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: AST/ALT =< 2.5 x upper limit of normal (ULN)
* PREVIOUSLY TREATED BORDERLINE RESECTABLE PDAC COHORT: Hemoglobin >= 8.0 mg/dL
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Pathologically proven adenocarcinoma of the pancreas by cytology or biopsy
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Confirmation of clinical stage of locally advanced
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: No prior chemotherapy or radiation therapy for PDAC
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Pregnancy and Nursing Status: Not pregnant and not nursing, For women of childbearing potential, a negative urine or blood pregnancy test done ≤ 7 days prior to registration is required
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Life expectancy greater than 6 months
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: ECOG performance status 0 or 1
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Absolute neutrophil count (ANC) >= 1,500/mm^3
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Platelet count >= 100,000/mm^3
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Creatinine =< 1.5 x upper limit of normal (ULN)
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Calc. creatinine clearance > 45 mL/min
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Total bilirubin =< 2.0 mg/dL
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: AST/ALT =< 2.5 x upper limit of normal (ULN)
* TREATMENT NAIVE LOCALLY ADVANCED PDAC COHORT: Hemoglobin >= 8.0 mg/dL
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Pathologically proven adenocarcinoma of the pancreas by cytology or biopsy
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Confirmation of clinical stage of locally advanced
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Prior chemotherapy for PDAC is allowed, as long as the regimen is considered a standard regimen for PDAC (e.g., gemcitabine, gemcitabine-cisplatin, gemcitabine/nab-paclitaxel, gemcitabine/capecitabine, FOLFIRINOX). This should be discussed with the study PIs prior to enrollment to ensure the regimen for a given patient is acceptable
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: No current use of immunosuppressive medication
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Not pregnant and not nursing, For women of childbearing potential, a negative urine or blood pregnancy test done =< 7 days prior to registration is required
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Life expectancy greater than 6 months
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: ECOG performance status 0 or 1
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Absolute neutrophil count (ANC) >= 1,500/mm^3
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Platelet count >= 100,000/mm^3
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Creatinine =< 1.5 x upper limit of normal (ULN)
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Calc. creatinine clearance > 45 mL/min
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Total bilirubin =< 2.0 mg/dL
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: AST/ALT =< 2.5 x upper limit of normal (ULN)
* PREVIOUSLY TREATED LOCALLY ADVANCED PDAC COHORT: Hemoglobin >= 8.0 mg/dL

Exclusion Criteria:

* TREATMENT NAIVE RESECTABLE PDAC COHORT: Previous treatment for PDAC with chemotherapy or radiation
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Active malignancy, except basal cell carcinoma
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Staging other than resectable PDAC
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Known uncontrolled (grade >=2) or active gastric or duodenal ulcer disease within 30 days of enrollment
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Prior surgical resection of pancreatic tumor
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Known contraindication to iodine-based or gadolinium-based intravenous (IV) contrast
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes, second or third degree atrioventricular heart block without a permanent pacemaker in place)
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Class III or IV congestive heart failure as defined by the New York Heart Association functional classification system < 6 months prior to screening
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Known active, uncontrolled (high viral load) human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection

  * Patients who have been vaccinated for hepatitis B and do not have a history of infection are eligible
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Female patients who are pregnant of breastfeeding
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Women of child-bearing potential and their male partners who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period. Acceptable methods of contraception are those that, alone or in combination, result in a failure rate of < 1% per year when used consistently and correctly
* TREATMENT NAIVE RESECTABLE PDAC COHORT: Have significant psychiatric, social, or medical condition(s) that could increase the subject's risk, interfere with protocol adherence, or affect the subject's ability to give informed consent
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: The patient is treatment naive
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: The patient previously received radiation to the abdomen for any reason
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Active malignancy, except basal cell carcinoma
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Staging other than resectable PDAC at the time of diagnosis
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Receiving any approved or investigational anti-neoplastic agent other than the chemotherapies specified in this protocol
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Known uncontrolled (grade >= 2) or active gastric or duodenal ulcer disease within 30 days of enrollment
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Prior surgical resection of pancreatic tumor
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Known contraindication to iodine-based or gadolinium-based IV contrast
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes, second or third degree atrioventricular heart block without a permanent pacemaker in place)
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Class III or IV congestive heart failure as defined by the New York Heart Association functional classification system < 6 months prior to screening
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Known active, uncontrolled (high viral load) HIV, hepatitis B or hepatitis C infection

  * Patients who have been vaccinated for hepatitis B and do not have a history of infection are eligible
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Female patients who are pregnant of breastfeeding
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Women of child-bearing potential and their male partners who are unwilling or unable to use an acceptable method of birth control to avoid pregnancy for the entire study period. Acceptable methods of contraception are those that, alone or in combination, result in a failure rate of < 1% per year when used consistently and correctly
* PREVIOUSLY TREATED RESECTABLE PDAC COHORT: Have significant psychiatric, social, or medical condition(s) that could increase the subject's risk, interfere with protocol adherence, or affect the subject's ability to give informed consent
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Previous treatment for PDAC with chemotherapy or radiation
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Active malignancy, except basal cell carcinoma
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Staging other than borderline resectable PDAC
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Known uncontrolled (grade >= 2) or active gastric or duodenal ulcer disease within 30 days of enrollment
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Prior surgical resection of pancreatic tumor
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Known contraindication to iodine-based or gadolinium-based IV contrast
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes, second or third degree atrioventricular heart block without a permanent pacemaker in place)
* TREATMENT NAIVE BORDERLINE RESECTABLE PDAC COHORT: Class III or IV congestive hea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2027-04-06 (Estimated); Study Completion 2027-04-06 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate | 12 weeks
  Major pathological response is any patient who has grade I or II treatment response. Grade I - 0% residual tumor cells in the specimen (pathologic complete response, grade II - 1 to < 5% residual tumor cells in the specimen.
Disease control rate | 6 months
  Measured as the proportion of patients without progression.

SECONDARY OUTCOMES:
Progression free survival | From the date of treatment initiation to the date of disease progression, recurrence after surgery or death from any cause whichever occurs first, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method. Comparisons of these time-to-event endpoints by important covariate subgroups will be made using the log-rank tests. Cox proportional hazards regression models will be explored to evaluate the associations between the time-to-event endpoints and covariates of interest.
Overall survival | From treatment start till death or last follow-up if the patient is alive, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method. Comparisons of these time-to-event endpoints by important covariate subgroups will be made using the log-rank tests. Cox proportional hazards regression models will be explored to evaluate the associations between the time-to-event endpoints and covariates of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene J Koay, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Douglas JE, Liu S, Ma J, Wolff RA, Pant S, Maitra A, Tamm EP, Bhosale P, Katz MHG, Varadhachary GR, Koay EJ. PIONEER-Panc: a platform trial for phase II randomized investigations of new and emerging therapies for localized pancreatic cancer. BMC Cancer. 2022 Jan 3;22(1):14. doi: 10.1186/s12885-021-09095-7. PMID 34980020
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT04481204/ICF_000.pdf